CLINICAL TRIAL: NCT07243704
Title: Reducing the Burden of Cardiovascular Events With Antiplatelet Therapy in Patients With IntraCerebral Haemorrhage.
Acronym: BEAT-ICH
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Christian Medical College and Hospital, Ludhiana, India (Other)
Collaborators: Indian Council of Medical Research (Other Government); St. Stephen's Hospital, Delhi (Other); Amrita Institute of Medical Sciences & Research Center (Other); Kasturba Medical College (Other); Bangur Institute of Neurosciences Kolkata (Unknown); Baptist Christian Hospital, Tezpur, India (Unknown); Christian Medical College, Vellore, India (Other); Lalitha Super Specialities Hospital (Other); Dr. Ramesh Cardiac and Multispecialty Hospital Guntur, India (Unknown); Government General Hospital Guntur, India (Unknown); Institute of Medical Sciences of the Banaras Hindu University, India (Other); All India Institute of Medical Sciences, Bhubaneswar (Other); KLE'S Dr Prabhakar Kore Hospital & MRC Balgaum (Unknown); Guru Gobind Singh Medical College & Hospital (Other); PBM Hospital Bikaner, India (Unknown); Excelcare Hospitals Guwahati (Unknown); Bharati Vidyapeeth DTU Medical College Pune, India (Unknown); All India Institute of Medical Sciences, Bilaspur (Unknown); KG Hospital and Post Graduate Medical Institute Coimbatore, India (Unknown); Tirunelveli Medical College, Tirunelveli, India (Unknown); Santokba Durlabhji Memorial Hospital (Other); Institute of Human Behaviour and Allied Sciences Delhi (Unknown); Government Medical College Trivandrum, India (Unknown); Jaiswal Multispeciality Hospital And Neuro Institute, Kota (Unknown); Shri Maharaja Hari Singh Hospital (Other Government); Government Medical College, Anantnag, India (Unknown); Narayana Medical College & Hospital (Other); Renova Institute of Neurological Sciences (RINS); Renova Century Hospital Hyderabad (Unknown); Rangaraya Medical College (Other); All India Institute of Medical Sciences, Raebareli, UP (Unknown); All India Institute of Medical Science, Patna, Bihar, India (Unknown); Sri Balaji Institute of Medical Sciences, Raipur, Chhattisgarh, India (Unknown); Manipal Group of Hospitals (Eastern Region), Kolkata, India (Unknown); Sree Chitra Tirunal Institute for Medical Sciences & Technology (Other Government); All India Institute of Medical Science, Guwahati (Unknown); All India Institute of Medical Science, New Delhi (Unknown); King George's Medical University, Lucknow, India (Unknown); P. D. Hinduja Hospital and Medical Research Centre (Unknown); KIMS-SUNSHINE Hospital, Hyderabad, India (Unknown); Sahyadri Superspeciality Hospital, Nasik (Unknown); Rajendra Institute of Medical Sciences, Ranchi, Jharkhand, India (Unknown)
Responsible Party: Principal Investigator, Jeyaraj D Pandian, Principal and Professor, Department of Neurology, Christian Medical College and Hospital, Ludhiana, India
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BEAT ICH
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Intracerebral Haemorrhage
Keywords: stroke; Intracerebral Haemorrhage; antiplatelet; Major adverse cardiovascular and cerebrovascular events; Randomized control trial; Secondary Prevention; Recurrent stroke
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin 75 mg OD (Active Comparator): The intervention is oral daily Aspirin 75 mg OD (antiplatelet drug monotherapy) in addition to standard care for secondary prevention after ICH based on the universal guidelines.
  Interventions: Drug: Aspirin 75 mg daily
- Placebo (Placebo Comparator): The control arm is placebo, which will be look-alike both as kits and tablets and will be prescribed in the same way as Aspirin: OD along with the standard secondary prevention after ICH.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin 75 mg daily — The intervention is oral daily Aspirin 75 mg OD The duration of the medication and follow-up will vary based on the recruitment timeline. If recruited during the first year of the trial, the first patient will take the medication for 2.5 years, and the last patient will get the IP for a minimum of 6 months.
  Other Names: Aspirin
  Arms: Aspirin 75 mg OD
Drug: Placebo — The intervention is a placebo to be taken OD. The duration of the placebo and follow-up will vary based on the recruitment timeline. If recruited during the first year of the trial, the first patient will take the placebo for 2.5 years, and the last patient will get the placebo for a minimum of 6 months.
  Other Names: Placebo OD
  Arms: Placebo

SUMMARY:
BEAT ICH will be a pragmatic, randomised, placebo-controlled, blinded, superiority clinical trial aiming to recruit 5676 patients aged ≥18 years who survive ICH and assign them 1:1 to starting antiplatelet monotherapy (Aspirin 75 mg od) versus placebo for the entire duration of the trial for preventing MACE. Recruitment duration is for 2.5 years. The duration of the medication and follow-up will vary based on recruitment timeline. If recruited during the first year of the trial, the patient will take the medication for three years or until the trial ends or an event occurs, with a matching follow-up period. If recruited towards the end of the trial, he/she will take the medication for six months and be followed up for the same duration. The trial's follow-up duration is three years. The patients will be recruited for 2.5 years, and the last recruit will have a minimum follow-up of six months. No new patients will be recruited within the last six months of the trial, but all the patients will be followed up until the end of the trial.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death and disability globally. Intracerebral haemorrhage (ICH) accounts for 10% to 15% of strokes in high-income countries and 20% to 50% in developing countries. The proportion of ICH ranges from 19% to 41% in India and is higher in Eastern India. Recurrent stroke rates are high worldwide; 15% in India (Kolkata), 41% in China, 6 and 13% in Taiwan.

ICH patients are at a risk of recurrent stroke (ICH and ischaemic) and other serious cardiovascular events, and yet there is no consensus regarding starting antiplatelet drugs for secondary prevention. RESTART is the only trial (pilot) that studied antiplatelet therapy and showed a decrease in recurrent ICH compared to no antiplatelet therapy, with a median follow-up of 2 years (IQR [1·0-3·0]). The recurrence rates were 4% in the intervention group versus 9% in the control group. There is no large stroke trial which has addressed this question.

Hence, plan is to initiate the BEAT-ICH trial, a randomized placebo-controlled trial of ICH patients where intervention arm patients will receive antiplatelet monotherapy (Aspirin 75mg) and the control arm will receive a placebo. The primary outcome will be determining whether antiplatelet monotherapy provides a net reduction in major adverse cardiovascular and cerebrovascular events (MACE) in the long term in ICH patients.

Trial Population:

This multi-centric study will be conducted at 50 stroke centres in India associated with the INSTRuCT Network. All patients presenting with symptoms of stroke to the hospital and admitted to the stroke units will be screened for eligibility and if met, will be included in the study. The BEAT ICH trial intends to recruit 5676 patients.

Study design:

Each site will have a team of neurologists (Principal Investigator and Co-Investigators) and a site coordinator. All ICH patients admitted to stroke and neurology wards, Outpatient department (OPD) or Inpatient Department (IPD) after 24 hrs to 3 months will be screened for eligibility by the image-conformed haemorrhagic stroke by the site neurologist.

Investigators will collect complete information about patients' demographics, comorbidities, functional status (US National Institutes of Health Stroke Scale score (NIHSS) and the modified Rankin Scale mRS)), previous antithrombotic therapy, medical history, medication history (at the time of stroke and at the time of randomisation), and intracerebral haemorrhage (image confirmed), vitals and assessments and hematoma details into a database via a secure web interface with in-built validation to ensure complete baseline data before randomisation.

Each patient will undergo brain imaging by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) as part of routine care at the time of ICH before enrolment. In case of any events, a second CT/MRI scan will be performed to assess for haematoma. All images will be saved in Digital Imaging and Communications in Medicine (DICOM) format and uploaded to the trial's Picture Archiving and Communication System (PACS) server.

After obtaining the consent form, Data will initially be recorded on paper case record forms (pCRF) and later entered into the electronic database. Patients not meeting the trial's eligibility criteria (screen failures) will also be captured in the database. All the recruited patients will be covered under comprehensive insurance for the entire trial duration. Randomisation will be initiated ≥24 hours after ICH onset up to 3 months, provided ICH growth has stopped by 24 hours after onset, followed by the investigational product (Aspirin/placebo) for the entire trial duration. All patients will receive additional standard care as per current gulidelines along with the intervention. Patients in the intervention arm will receive Aspirin 75 mg daily, and the control arm will receive a placebo tablet of similar shape, size, and colour daily. Both investigational products will be pills that look similar in appearance. Pharmaceutical company will centrally manufacture, label, and dispense the investigational products under the supervision of the pharmacologist at Christian Medical College and Hospital (CMCL). Since this trial is triple-blinded, the investigator, coordinator, and patient will be blinded to the allocated study treatment. Only the pharmacologist will decode in case of an event requiring a medication change in an emergency.

Each site will have a stock for a duration of one year, with new investigational products delivered yearly or based on prior consumption and follow-up requirements. Each site is expected to have a dedicated IP room for this purpose. Once delivered, the site will handle the storage, dispensing, and destruction of the investigational products, unused IP, and returned kits under the hospital's waste disposal management protocols with strict supervision.

The duration of the medication and follow-up will vary based on recruitment timeline. If recruited during the first year of the trial, the patient will take the medication for three years or until the trial ends or an event occurs, with a matching follow-up period. If recruited towards the end of the trial, he/she will take the medication for six months and be followed up for the same duration. The trial's total duration is three years. The patients will be recruited for 2.5 years, and the last recruit will have a minimum follow-up of six months. No new patients will be recruited within the last six months of the trial, but all the patients will be followed up until the end of the trial.

All patients will remain in the trial until the end of the study period (3 years to the max)/event/death/withdrawal. If a patient develops an event, the investigational product will be stopped, and treatment will be initiated based on the event and clinical guidelines. Unused investigational products will be returned to the site. If required, the trial pharmacologist will handle decoding after an event. Site research staff will capture all event-related data and submit it to the database and the site ethics committee for review. The central independent event adjudication committee will also review this data. In case of patient withdrawal or death, the investigational product will also be returned to the site. All patients will be analysed using the intention-to-treat principle, even if they withdraw at any point during the trial.

Patients will be called for face-to-face visits every 3 months to dispense the investigational product. Kits will be labelled as BEAT-ICH trial medication, with a unique kit number for identification for each patient. Each kit will contain 100 tablets, including a buffer of 10 tablets for delayed visits/buffer dose. The site coordinators will call the patient 15 days before the visit as a reminder to come to the hospital to take the next batch of IP. Monthly telephonic follow-ups will ensure medication adherence and detect events. Patients will be encouraged to report events during the interim follow-up period. At each visit, patients will return used kits and unused medication (expected return of approximately 10 tablets on every three-month visit) to monitor medication adherence.

The need for this study:

The BEAT-ICH trial has the potential to reduce the recurrent stroke rate and MACE after ICH. In addition, this trial will address the important question of the safety of antiplatelet use in ICH patients. If completed, this trial can change Clinical practice and guidelines globally, as aspirin is a low-cost drug that can be provided at all levels of healthcare in India.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* First-ever Intracerebral Haemorrhage
* Presenting ≥24 hrs up to 3 months of stroke symptoms confirmed by brain imaging
* CT /MRI confirming Intracerebral Haemorrhage
* Alive ≥24 hours after non-traumatic ICH

Exclusion Criteria:

* ICH is known to be due to trauma, a structural cause (e.g., aneurysm, arteriovenous malformation, cerebral cavernous malformation, venous thrombosis, or tumour), or haemorrhagic transformation of cerebral infarction
* Glasgow coma score ≤5
* Taking any antiplatelet or anticoagulant therapy 15 days prior to randomization.
* Women pregnant, breastfeeding, childbearing potential, and not using contraceptives
* Enrolled in any other clinical trial
* Sick or compromised patients with life expectancy of less than a year
* Geographical or other factors that prohibit long-term follow-up

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5676 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2029-02-14 (Estimated); Study Completion 2029-02-14 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | 3 years
  To reduce the risk of first MACE (stroke, myocardial infarction, hospitalisation, or death) with antiplatelet monotherapy in ICH patients. The components of the MACE include ischemic stroke, haemorrhagic stroke, hospitalisation due to stroke (ischemic, haemorrhagic, subarachnoid haemorrhage), myocardial infarction, coronary artery disease, cerebral and cardiovascular death due to any vascular causes (including pulmonary embolism, gastrointestinal haemorrhage) or death due to non-Cerebrovascular and cardiovascular causes.

SECONDARY OUTCOMES:
Major bleeding | 3 years
  To study the safety composite outcome of major bleeding (all major haemorrhagic events that are fatal or result in hospitalisation)
Medication adherence | 3 years (every 3 months) till study end
  To check the adherence of aspirin vs placebo.
modified Rankin Scale | 3 years (every 3 months) till study end
  To check the modified Rankin Scale (mRS), a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a ICH stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Jeyaraj D Pandian, MD, DM, Principal Investigator — Christian Medical College and Hospital, Ludhiana, Punjab, India
Locations (40):
- India (40):
  - Government General Hospital, Guntur, Andhra Pradesh
  - Lalitha Super Specialty Hospital, Guntur, Andhra Pradesh
  - Dr Ramesh Cardiac and Multispecialty Hospital, Guntur, Andhra Pradesh
  - Government General Hospital, Kākināda, Andhra Pradesh
  - Narayana Medical College and Hospital, Nellore, Andhra Pradesh
  - Apollo Excelcare Hospitals, Guwahati, Assam
  - Baptist Christian Hospital, Tezpur, Assam
  - All India Institute of Medical Science, Patna, Bihar
  - All India Institute of Medical Sciences, Bilāspur, Himachal Pradesh
  - Government Medical College, Anantnag, Jammu and Kashmir
  - Shri Maharaja Hari Singh (SMHS) Hospital, Srinagar, Jammu and Kashmir
  - Rajendra Institute of Medical Sciences, Ranchi, Jharkhand
  - KLE's Dr. Prabhakar Kore Hospital & Medical Research Centre, Belagavi, Karnataka
  - Kasturba Medical College Manipal, Manipal, Karnataka
  - Amrita Institute for Medical Sciences and Research Center, Kochi, Kerala
  - Government Medical College Trivandrum, Thiruvananthapuram, Kerala
  - Sree Chitra Tirunal Institute for Medical Sciences and Technology, Thiruvananthapuram, Kerala
  - P. D. Hinduja Hospital and Medical Research Centre, Mumbai, Maharashtra
  - Sahyadri Superspeciality Hospital, Nashik, Maharashtra
  - Bharati Vidyapeeth DTU Medical College, Pune, Maharashtra
  - Institute of Human Behaviour and Allied Sciences, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences, Bhubaneswar, Odisha
  - Guru Gobind Singh Medical College and Hospital, Farīdkot, Punjab
  - PBM Hospital, Bikaner, Rajasthan
  - Santokba Durlabhji Memorial Hospital, Jaipur, Rajasthan
  - Jaiswal Hospital and Neuro Institute, Kota, Rajasthan
  - KG Hospital and Post Graduate Medical Institute Coimbatore, Coimbatore, Tamil Nadu
  - Tirunelveli Medical College, Tirunelveli, Tamil Nadu
  - Christian Medical College Vellore, Vellore, Tamil Nadu
  - King George's Medical University, Lucknow, Uttar Pradesh
  - All India Institute of Medical Sciences, Raebareli, Uttar Pradesh
  - Institute of Medical Sciences of the Banaras Hindu University (BHU), Varanasi, Uttar Pradesh
  - Bangur Institute of Neurosciences, Kolkata, West Bengal
  - St Stephen's Hospital, Delhi
  - All India Institute of Medical Science, Guwahati
  - KIMS-Sunshine Hospitals, Hyderabad
  - Renova Institute of Neurological Sciences (RINS); Renova Century Hospital, Hyderabad
  - Manipal Group of Hospitals (Eastern Region), Kolkata
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow
  - All India Institute of Medical Science, New Delhi

IPD SHARING:
Plan to Share IPD: No
All information collected from medical records for the study will be stored electronically in a specifically designed database at the Christian Medical College and Hospital, Ludhiana, Punjab, India. Participants information will be identified only by their initials and a study registration number. Any information transferred electronically will be coded to protect confidentiality. All computer records will be password-protected. The study results may be presented at conferences or in scientific publications, but individual participants will not be identifiable. If needed, data will be available in future for other researchers outside the primary research group for secondary purposes, such as metaanalyses, reanalysis, or replication of results.

REFERENCES:
- [Background] RESTART Collaboration. Effects of antiplatelet therapy after stroke due to intracerebral haemorrhage (RESTART): a randomised, open-label trial. Lancet. 2019 Jun 29;393(10191):2613-2623. doi: 10.1016/S0140-6736(19)30840-2. Epub 2019 May 22. PMID 31128924
- [Background] Wong YS, Tsai CF, Ong CT. Risk factors for stroke recurrence in patients with hemorrhagic stroke. Sci Rep. 2022 Oct 13;12(1):17151. doi: 10.1038/s41598-022-22090-7. PMID 36229641
- [Background] Katan M, Luft A. Global Burden of Stroke. Semin Neurol. 2018 Apr;38(2):208-211. doi: 10.1055/s-0038-1649503. Epub 2018 May 23. PMID 29791947
- [Background] Banerjee TK, Das SK. Fifty years of stroke researches in India. Ann Indian Acad Neurol. 2016 Jan-Mar;19(1):1-8. doi: 10.4103/0972-2327.168631. PMID 27011621